CLINICAL TRIAL: NCT05282225
Title: Adaptive Intervention to Prevent Adolescent Suicidal Behavior Following Psychiatric Hospitalization
Brief Title: Adaptive Intervention for Adolescents Following Inpatient Psychiatric Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ewa Czyz, Assistant Professor, Department of Psychiatry, University of Michigan, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HUM00204329; 1R01MH126871 (NIH)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Suicide; Suicide, Attempted; Suicidal Ideation; Self Harm
Keywords: Adaptive Intervention; Technology-based interventions; In-patient; Sequential, Multiple Assignment, Randomized Trial (SMART); Adolescent; Safety planning; Mobile technology
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicidal Ideation; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Sequential, multiple assignment, randomized trial (SMART) design of an adjunctive, multi-component intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- MI-SP +supportive Texts + monitoring (Sequence A) (Experimental): Sequencing of intervention components (Phase 1 and Phase 2) resulting in Sequence or Group A: Participants will receive the in-person MI-enhanced safety plan (MI-SP) during hospitalization followed by 4 weeks of supportive Texts and monitoring post discharge.
  Interventions: Behavioral: MI- Safety Plan; Behavioral: Texts messages; Behavioral: Monitoring
- MI-SP + monitoring (Sequence D) (Experimental): Sequencing of intervention components (Phase 1 and Phase 2) resulting in Sequence or Group D: Participants will receive the in-person MI-enhanced safety plan (MI-SP) during hospitalization followed by 4 weeks of monitoring post discharge.
  Interventions: Behavioral: MI- Safety Plan; Behavioral: Monitoring
- MI-SP + supportive Texts + monitoring + portal follow-up for non-responders (Sequence B). (Experimental): Sequencing of intervention components (Phase 1 and Phase 2) resulting in Sequence or Group B: Participants will receive the in-person MI-enhanced safety plan (MI-SP) during hospitalization followed by 4 weeks of supportive Texts and monitoring post discharge in addition to the portal follow-up for non-responders.
  Interventions: Behavioral: MI- Safety Plan; Behavioral: Texts messages; Behavioral: Monitoring; Behavioral: Portal follow-up
- MI-SP + supportive Texts + monitoring + booster call for non-responders (Sequence C) (Experimental): Sequencing of intervention components (Phase 1 and Phase 2) resulting in Sequence or Group C: Participants will receive the in-person MI-enhanced safety plan (MI-SP) during hospitalization followed by 4 weeks of supportive Texts and monitoring post discharge in addition to the booster call for non-responders.
  Interventions: Behavioral: MI- Safety Plan; Behavioral: Texts messages; Behavioral: Monitoring; Behavioral: Booster call
- MI-SP + monitoring + portal follow-up for non-responders (Sequence E) (Experimental): Sequencing of intervention components (Phase 1 and Phase 2) resulting in Sequence or Group E: Participants will receive the in-person MI-enhanced safety plan (MI-SP) during hospitalization followed by 4 weeks of monitoring post discharge in addition to the portal follow-up for non-responders.
  Interventions: Behavioral: MI- Safety Plan; Behavioral: Monitoring; Behavioral: Portal follow-up
- MI-SP + monitoring + booster call for non-responders (Sequence F) (Experimental): Sequencing of intervention components (Phase 1 and Phase 2) resulting in Sequence or Group F: Participants will receive the in-person MI-enhanced safety plan (MI-SP) during hospitalization followed by 4 weeks of monitoring post discharge in addition to the booster call for non-responders.
  Interventions: Behavioral: MI- Safety Plan; Behavioral: Monitoring; Behavioral: Booster call

INTERVENTIONS:
Behavioral: MI- Safety Plan — The MI-enhanced safety plan (MI-SP) component is delivered during hospitalization and includes an individual and family meetings. The goal of the individual meeting with the adolescent is to develop an individualized safety plan for use during a suicidal crisis. This "best practices" approach of safety planning is augmented with Motivational Interviewing (MI) as a core strategy to explicitly elicit adolescents' motivation and commitment to behavior change (i.e. use safety plan; adaptive coping), address barriers or ambivalence, and strengthen self-efficacy. The focus of the family meeting, which is similarly guided by MI, is to prepare parents/guardians, with input from the adolescent, for how they may support the adolescent in implementing the individualized safety plan after discharge and on strengthening parents' commitment and self-efficacy
Behavioral: Texts messages — For participants randomized to receive supportive text messages (Texts), text messages will be sent daily for 4 weeks. The messages will be tailored to encourage use of individualized coping strategies identified as part of safety planning at hospitalization and will include additional adaptive coping tools and resources. The text message content and tone will be consistent with principles of MI.
  Arms: MI-SP + supportive Texts + monitoring + booster call for non-responders (Sequence C); MI-SP + supportive Texts + monitoring + portal follow-up for non-responders (Sequence B).; MI-SP +supportive Texts + monitoring (Sequence A)
Behavioral: Monitoring — Adolescent participants will complete daily surveys for 4 weeks (including assessment of suicidal ideation, behavior, and other relevant risk and protective factors) and these will be monitored daily to identify presence of heightened suicidal ideation and presence of suicidal behavior. In addition, daily surveys will be used to determine if adolescents are sufficient responders to Phase 1 intervention.
Behavioral: Portal follow-up — This will be part of Phase 2. The portal follow-up will similarly address content offered in the booster call. For the adolescent, the focus will be on revisiting and adjusting the safety plan, addressing barriers to safety plan adherence, as well as enhancing motivation and self-efficacy to use healthy coping. For the parent, portal communication will focus on revisiting safety recommendations provided as part of MI-SP, addressing barriers in implementing safety recommendations and in supporting the adolescent's safety plan use, as well as enhancing parents' motivation and self-efficacy in these areas. The portal will enable additional asynchronous contacts up to 3 weeks to provide added support and problem solving, based on identified barriers and concerns, to promote post-discharge behavior change. Counselors will initiate approximately 6 contacts with adolescents and, separately, with parents over 3 weeks as soon as non-response is detected.
  Arms: MI-SP + monitoring + portal follow-up for non-responders (Sequence E); MI-SP + supportive Texts + monitoring + portal follow-up for non-responders (Sequence B).
Behavioral: Booster call — The focus of the post-discharge booster phone call with adolescent and with parent, each conducted separately, is to further adjust the safety plan to better meet post-discharge needs, to further enhance adolescents' motivation and commitment to use coping strategies, and to further support adolescents' and parents' self-efficacy to manage suicidal crises.
  Arms: MI-SP + monitoring + booster call for non-responders (Sequence F); MI-SP + supportive Texts + monitoring + booster call for non-responders (Sequence C)

SUMMARY:
This study is being completed to examine different combinations of technology-augmented strategies to identify an effective Adaptive intervention (AI) addressing post-discharge suicide risk with high implementation potential.

DETAILED DESCRIPTION:
The proposed study is a sequential multiple assignment randomized trial (SMART) to identify an effective adaptive intervention (AI) for adolescents at elevated suicide risk transitioning from acute psychiatric care. Participants will be initially randomized to Motivational Interview (MI)-enhanced safety planning (MI-SP) or to MI-SP with supportive text messages delivered for four weeks after discharge (Texts) (Phase 1 intervention). Adolescents who are classified as Phase 1 non-responders at the end of the first or at the end of the second week post-discharge, based on their responses to daily surveys , will be re-randomized to either added booster call or portal follow-up (Phase 2 intervention). Those classified as Phase 1 responders at the end of the second week post discharge will continue with the initially assigned intervention options. Thus, participants will receive one of six treatment sequences resulting from the different intervention components or their combinations. These six treatment sequences, in turn, will form four AIs.

The study team anticipates that AIs that begin with MI-SP plus text-based support will have:

* lower odds of suicidal behavior 3 months post discharge
* longer time to suicidal behavior over the 6 month follow-up
* less severe suicidal ideation over the 6-month follow-up

Additionally, the study team anticipates that the AI that begins with MI-SP + Texts followed by portal follow-up for non-responders will lead to:

* lowest odds of suicidal behavior within 3 months
* longest time to suicidal behavior over the 6 month follow up
* least severe ideation over the 6-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* A suicide attempt in the last month or (2) past-week suicidal ideation (based on the Columbia-Suicide Severity Rating Scale (C-SSRS). In the absence of C-SSRS ratings in the chart, attending physician indication in the chart of the presence of suicidal ideation within the last week or the presence of a suicide attempt in the last month will be used.

Exclusion Criteria:

* Adolescent presenting with severe cognitive impairment or with altered mental status (acute psychosis or acute manic state)
* Transfer to medical unit or residential placement
* No availability of a legal guardian
* Adolescent not owning a cell phone.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The Columbia-Suicide Severity Rating Scale (C-SSRS) | up to 3 months after discharge
  This is a semi-structured interview and will be used to assess suicidal behavior (actual, interrupted, aborted suicide attempts).

SECONDARY OUTCOMES:
C-SSRS will be used to assess the secondary outcome of time-to-suicidal behavior within 6 months of discharge | up to 6 months
  The Columbia-Suicide Severity Rating Scale (C-SSRS), a semi-structured interview, will be used to assess suicidal behavior (actual, interrupted, aborted suicide attempts).
Suicidal Ideation Questionnaire-Junior (SIQ-JR) | up to 6 months after discharge
  Suicide ideation will be measured using the Suicidal Ideation Questionnaire (SIQ-JR), a 15-item measure of adolescents' distress and suicidal intent. Scale scores range from 0 to 90, with higher scores meaning a worse outcome (i.e., greater suicide ideation).

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Czyz, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of Michigan's (Child and Adolescent Psychiatric Inpatient Program), Ann Arbor, Michigan
  - Henry Ford Health System (Kingwood Hospital), Detroit, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No